CLINICAL TRIAL: NCT00705120
Title: Treatment of Severe (Types II and III) Osteogenesis Imperfecta by Allogeneic Bone Marrow Transplantation
Brief Title: Treatment of Severe Osteogenesis Imperfecta by Allogeneic Bone Marrow Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Edwin M Horwitz, MD, PhD, St. Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOIT
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2008-06-25 (Estimated); Status verified 2008-06

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis Imperfecta; Bone Marrow Cell Transplantation; Mesenchymal Stem Cells; Stem Cell Transplantation, Mesenchymal
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Bone Marrow Transplantation; Whole-Body Irradiation; Cyclophosphamide; Cyclosporine; Mesenchymal Stem Cell Transplantation; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other)
  Interventions: Other: Bone Marrow Cell Transplantation; Drug: Cyclophosphamide; Drug: Cyclosporin; Procedure: Mesenchymal Stem Cell Transplantation; Drug: Busulfan
- 2 (Other)
  Interventions: Other: Bone Marrow Cell Transplantation; Radiation: Irradiation, Total Body; Drug: Cyclophosphamide; Procedure: Mesenchymal Stem Cell Transplantation; Drug: Busulfan

INTERVENTIONS:
Other: Bone Marrow Cell Transplantation
Radiation: Irradiation, Total Body
  Arms: 2
Drug: Cyclophosphamide
Drug: Cyclosporin
  Arms: 1
Procedure: Mesenchymal Stem Cell Transplantation
Drug: Busulfan

SUMMARY:
This protocol was a prospective, Phase I study of allogeneic bone marrow transplantation (BMT) as the primary therapy for Osteogenesis Imperfecta Types II and III. Compatible sibling donors and unrelated donors were stratified and analyzed according to the type of donor. All patients with a sibling donor will received a chemotherapy conditioning regimen; a non-T cell depleted allogeneic marrow, and GVHD prophylaxis. All patients with an unrelated donor will receive a chemoradiotherapy conditioning regimen, a T-cell depleted allogeneic marrow, and GVHD prophylaxis. The primary objective of this study was to investigate the safety and toxicity of these BMT procedures in this particular population.

DETAILED DESCRIPTION:
The secondary objective of the protocol assessed the engraftment of donor mesenchymal cells and their ability to increase the synthesis of normal type I procollagen relative to the synthesis of mutated type I procollagen and to assess whether BMT improves the bone structure and the clinical condition of these patients with OI.

ELIGIBILITY:
Inclusion Criteria:

* Patient has diagnosis of OI Type II or III. Because there are no specific, defined clinical criteria consistently used to make this diagnosis, we provide the following clinical guidelines to assist in diagnosis. Any appropriate combinations of the following clinical findings will be acceptable.

Diagnosis of OI Type II

* Antenatal ultrasonography (if performed for other indications) by established obstetric impressions including short femurs, a small thoracic cage and poorly mineralized bones. Analysis of collagen synthesized from cultured cells obtained from chorionic villus sampling (CVS) may establish the diagnosis; however, no CVS will be performed specifically for enrollment into this study.
* Clinical examination including prematurity, low birth weight, characteristic facies (blue sclera, beaked nose, extremely soft calvarium), "frog-leg" hips, small thoracic cavity, fractures at birth or shortly thereafter, loose skin or lax joints that cannot be readily explained by other factors.
* Radiographic evaluation demonstrating various aspects of the characteristic picture of telescoped femur, bowed tibias, beaded ribs, flattened vertebral bodies and virtual absence of calvarial mineralization.

Diagnosis of OI Type III

* Antenatal ultrasonography (performed for other indications) by established obstetric impressions for this more moderate form of OI. Chorionic villus sampling will be accepted as above.
* Clinical examination including short stature, bony deformities, many fractures at birth or shortly thereafter. Blue scleras and dental abnormalities are also common.
* Radiographic abnormalities including thin, osteopenic bones of the limbs with evidence of fractures, growth plate abnormalities, and an undermineralized calvarium.
* Diagnosis of other diseases with possibly similar presentation to OI (e.g. hypophosphatasia and rickets) should be excluded by obtaining a serum calcium, phosphate and alkaline phosphatase. These parameters can be expected to be within normal limits (alkaline phosphatase may be somewhat elevated) in patients with OI.
* Age less than 3 years at time of transplant.
* Parents or legal guardians must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side effects, including treatment related mortality. Patients or their guardians will be given a copy of the consent form.
* Identification of a suitable bone marrow donor.
* Any donor must be of sufficient size so that adequate bone marrow may be harvested.
* HLA mismatched sibling or unrelated donor. DNA typing will be per- formed on unrelated donors. Donors must be a 6/6 match or a 5/6 match (with serologic mismatch at a single Class I allele or mismatch at a single DR1 allele).

Exclusion Criteria:

* Patients who are ventilatory dependent due to primary lung parenchymal disease prior to BMT.
* Patients with evidence of basilar invagination/compression.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 1995-11; Primary Completion 2000-07 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and toxicity of allogeneic bone marrow transplantation (BMT) in children with severe Osteogenesis Imperfecta (OI) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kasow, DO, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: Related Info — http://www.stjude.org